CLINICAL TRIAL: NCT01149707
Title: A 2-Week Exploratory Randomized, Double-Blind, Parallel-Group, Dose-Ranging, Placebo-Controlled Safety, Tolerability, Biomarker and Efficacy Clinical Study of PUR 0110 Rectal Enema in Mild-to-Moderate Distal Ulcerative Colitis
Brief Title: Safety, Tolerability, Efficacy Study of PUR 0110 Rectal Enema in Mild-to-Moderate Distal Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PurGenesis Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG09 PUR 0210 002; 2009 017839 18 (EudraCT Number); 29PS1617 (Other: FOCUS Clinical Drug Development GmbH)
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Left-Sided Ulcerative Colitis; Proctosigmoiditis
Keywords: PUR 0110; PUR 0110 Rectal Enema; Distal Ulcerative Colitis; Left-Sided Ulcerative Colitis; Mild; Moderate
MeSH Terms: conditions — Proctocolitis; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PUR 0110 Rectal Enema 250 mg (Experimental): Active treatment
  Interventions: Drug: PUR 0110 Rectal Enema 250 mg
- PUR 0110 Rectal Enema 500 mg (Experimental): Active treatment
  Interventions: Drug: PUR 0110 Rectal Enema 500 mg
- PUR 0110 Rectal Enema 1000 mg (Experimental): Active treatment
  Interventions: Drug: PUR 0110 Rectal Enema 1000 mg
- Placebo Enema (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo Enema

INTERVENTIONS:
Drug: PUR 0110 Rectal Enema 250 mg — PUR 0110 Rectal Enema 250 mg, once-daily, intrarectally
  Other Names: Active treatment arm
  Arms: PUR 0110 Rectal Enema 250 mg
Drug: PUR 0110 Rectal Enema 500 mg — PUR 0110 Rectal Enema 500 mg, once-daily, intrarectally
  Other Names: Active treatment arm
  Arms: PUR 0110 Rectal Enema 500 mg
Drug: PUR 0110 Rectal Enema 1000 mg — PUR 0110 Rectal Enema 1000 mg, once-daily, intrarectally
  Other Names: Active treatment arm
  Arms: PUR 0110 Rectal Enema 1000 mg
Drug: Placebo Enema — Placebo Enema, once-daily, intrarectally
  Other Names: Placebo arm
  Arms: Placebo Enema

SUMMARY:
PUR 0110 is a 100% natural novel investigational medicinal product that has been demonstrated in several in vitro and in vivo pharmacology studies to have potent anti-inflammatory, anti-oxidative and immunomodulatory effects. This exploratory Phase 2a study is a first-in-patient study to evaluate the safety, tolerability, biomarker effect and efficacy of PUR 0110 rectal enema in patients with active mild-to-moderate distal ulcerative colitis (UC).

The study is a multicenter, randomized, double-blind, parallel-group, dose-ranging, placebo-controlled study. To be eligible for inclusion into the study, patients must either be newly diagnosed or have on-going active mild-to-moderate distal ulcerative colitis of at least 3 months duration confirmed in either case by flexible sigmoidoscopy and biopsy at the Screening Visit. In addition, patients must have a modified Mayo score of ≥5 to ≤10 including a sigmoidoscopy inflammation grade and rectal bleeding scores of ≥2 each. Eligible patients will be randomly assigned to receive either PUR 0110 250 mg, 500 mg or 1000 mg or placebo rectal enema in a 1:1:1:1 ratio. Patients will self-administer the assigned study medication intrarectally once-daily at bedtime (10:00 p.m +/- 1 hour) for 2 weeks.

Patients will be evaluated for safety by adverse events, clinical laboratory tests, vital signs, physical examination, electrocardiogram (ECG), and concomitant medications. Efficacy evaluations will include the modified Mayo score, patient-defined response and remission, Investigator Assessment of Ulcerative Colitis Symptom Score, Inflammatory Bowel Disease Questionnaire (IBDQ), and biomarkers of inflammation, apoptosis and total cell death, lipid peroxidation and in vivo oxidative stress, and antioxidant defense mechanisms in plasma, serum, urine, feces and biopsy tissue. Patients will have a flexible sigmoidoscopy and biopsy 12 hours after the last dose of study medication.

DETAILED DESCRIPTION:
Safety/Primary Outcome Parameters:

* Incidence, nature and severity of adverse events
* Incidence, nature and severity of clinical laboratory test abnormalities

Efficacy/Secondary Outcome Parameters:

* Clinical remission defined as an endoscopy score of ≤ 1, a rectal bleeding score of 0, and an improvement or no change from baseline in the stool frequency score at the end of 2 weeks of treatment / withdrawal visit;
* Clinical response rate defined as the percentage of patients with a drop of ≥3 points from the baseline overall modified Mayo score;
* Patient defined response and remission rates;
* Change from baseline in the overall modified Mayo score (Disease Activity Index);
* Change from baseline in each of the 4 individual sub-scores of the modified Mayo score;
* Change from baseline in Investigator Assessment of UC Symptom Score (total and individual symptom scores)
* Change from baseline in IBDQ score (total and the 4 individual dimension scores)
* Proportion of patients with treatment failure;
* Change from baseline in serum lutein levels;
* Change from baseline in C-reactive protein (CRP), high sensitivity CRP (hs-CRP), erythrocyte sedimentation rate (ESR), fecal calprotectin (FCP), and fecal lactoferrin (FL).
* Change from baseline in exploratory biomarkers including: serum interleukin-2 (IL-2), IL-6, IL-8, interferon-gamma (IFN-gamma), tumor necrosis factor-alpha (TNF-α), transforming growth factor-beta (TGF-beta), IL-4, IL-10, IL-17, IL-23, human beta-Defensin-2 (hBD-2), malondialdehyde (MDA), lipoxin A4 (LXA4), glutathione (GSH), M30 and M65 apoptosomes in serum and biopsies, and plasma and urinary isoprostane levels.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient males and females between 18 and 75 years.
2. Females of child bearing potential must have a negative serum pregnancy test (beta-human chorionic gonadotropin) at screening and must be sexually inactive (abstinent) for 3 months prior to dosing and throughout the study or be using one of the following acceptable methods of contraception:

   * barrier methods (condom, diaphragm with spermicide);
   * Intrauterine device (IUD) in place for at least 3 months;
   * surgical sterilization of the partner (vasectomy for at least 6 months); or
   * hormonal contraceptives for at least 3 months prior to dosing. [Female subjects of childbearing potential must be advised to remain sexually inactive or maintain the same method of contraception for ≥7 days following the end of dosing of study treatment]
3. Patients newly diagnosed or with ongoing active distal ulcerative colitis of >3 months duration, confirmed by flexible sigmoidoscopy during screening, and extending 5 to 50 cm from the anal margin. Sigmoidoscopy must be conducted within not more than 3 +/- 1 days before the Baseline (Day 0) Visit.
4. Patients with ongoing active distal ulcerative colitis of ≥3 months duration must be on a stable dose of oral mesalamine (5-ASA) for ≥2 months before the Baseline (Day 0) Visit.
5. Modified Mayo Score (Disease Activity Index) of ≥5 to ≤10 at Baseline, including a sigmoidoscopic inflammation grade score of ≥2 and a rectal bleeding score ≥2.
6. Negative stool test at screening to rule out parasites, bacterial pathogens and Clostridium difficile.
7. Able and willing to fill in (maintain) daily diary cards from Day -7 to Day 21 of the study.
8. Able to provide voluntary written informed consent prior to initiation of screening, must be capable of following the verbal and written study instructions, and be able to commit to the return visits during the entire period of the study.

Exclusion Criteria:

1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatological, neurological, or psychiatric disease, that could compromise patient's ability to participate in the study, and/or interfere with absorption of the study drug or the interpretation of the study data.
2. Patients with a diagnosis of Crohn's disease.
3. Patients with a modified Mayo score of ≥11 at the Screening (Day -7 & Day -3) Visits.
4. Patients at immediate or significant risk of toxic megacolon; those with bowel stricture, colonic dysplasia, adenoma or carcinoma.
5. Use of botanical treatments and supplements for ulcerative colitis within 14 days prior to the Baseline Visit.
6. Patients with any enteric pathogens, ova or parasites, or Clostridium difficile toxin in stool.
7. Female patients with a positive pregnancy test or lactating at the Screening/Baseline Visits.
8. History of allergic reaction or hypersensitivity to spinach, spinach tablet, spinach powder or spinach extract; and to latex, molds and mushrooms.
9. History of gout, pseudogout or hyperuricemia, or kidney stones.
10. History of pseudoallergic hypersensitivity to the food color additives, tartrazine (E102), sunset yellow (E110) and FD & C Blue No.1 (Brilliant blue FCF; E133), allergic asthma, aspirin intolerance, and severe or multiple allergies.
11. Past medical history of significant gastrointestinal surgery including but not limited to colostomy, ileostomy, or previous colonic surgery other than appendectomy.
12. Patients with anatomical abnormalities of the colon, e.g., short bowel or other abnormalities.
13. Patients with any current infectious, ischemic, or immunologic disease with gastrointestinal involvement.
14. Patients with a history of failure to retain enemas.
15. Use of antibiotics for reasons related to the primary diagnosis or for other gastrointestinal-related conditions within 14 days of Baseline Visit.
16. Patients who used non-steroidal anti-inflammatory drugs (NSAIDs), including cyclooxygenase-2 (COX-2) inhibitors, within 14 days prior to Baseline Visit. Except aspirin ≤325 mg/day for cardiovascular prophylaxis.
17. Patients who used the following medications used for treating ulcerative colitis from the times indicated below to the end of Week 3 (Visit 6):

    * Topical intrarectal corticosteroids or topical intrarectal mesalamine within 14 days of Baseline Visit;
    * Systemic corticosteroids (oral or injectable, including adrenocorticotropic hormone [ACTH]) within 30 days of Baseline Visit;
    * Immunosuppressant therapy (methotrexate, azathioprine, 6-mercatopurine or cyclosporine) within 60 days of Baseline Visit; and
    * Biologic therapy (tumor necrosis factor-α inhibitors, monoclonal antibodies, etc.) within 90 days of Baseline Visit.
18. Patients with a history of active malignancy within the past 5 years except for squamous cell or basal cell cancers of the skin.
19. History of any clinical laboratory abnormality deemed significant by the Principal Investigator.
20. History of significant alcohol or drug abuse within one year prior to the Screening Visit.
21. Patients who tested positive at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg) or hepatitis C virus (HCV).
22. Exposure to any investigational or non-registered drug within 30 days prior to administration of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06-01; Primary Completion 2014-10-01 (Actual); Study Completion 2015-06-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events | At Week 2
  Safety & Tolerability of PUR0110 rectal enema compared to placebo as per Incidence, nature and severity of adverse events (AEs); and abnormal clinical laboratory test results.

SECONDARY OUTCOMES:
Effectiveness of PUR0110 on remission rate | At week 2
  Effectiveness of PUR0110 compared to placebo as per Clinical remission rate with clinical remission defined as an endoscopy score of ≤ 1, a rectal bleeding score of 0, and an improvement or no change from baseline in the stool frequency score at the end of 2 weeks of treatment / withdrawal visit.
Effectiveness of PUR0110 on clinical response rate | At week 2
  Effectiveness of PUR0110 compared to placebo as per : Clinical response rate defined as the percentage of subjects with a drop of ≥3 points from the baseline overall modified Mayo score.
Effectiveness of PUR0110 on subject response and remission rate | At week 2
  Effectiveness of PUR0110 compared to placebo as per Subject defined response and remission rates based on their well being : 1= much better; 2= some better; 3=a little better; 4= about the same; 5=a little worse; 6= some worse & 7= much worse.ed as : o= none; 1 = mild; 2=moderate, 3=severe and 4 = incapacitating.
Effectiveness of PUR0110 on overall Mayo score | At week 2
  Effectiveness of PUR0110 compared to placebo as per Change from baseline in the overall modified Mayo score.
Effectiveness of PUR0110 on in each of the 4 individual sub-scores of the modified Mayo score. | At week 2
  Effectiveness of PUR0110 compared to placebo as per Change from baseline in each of the 4 individual sub-scores of the modified Mayo score.
Effectiveness of PUR0110 on investigator assessment of ulcerative colitis symptom score | At week 2
  Effectiveness of PUR0110 compared to placebo as per Change from baseline in investigator assessment of ulcerative colitis symptom score : 0= none; 1= Mild; 2=Moderate; 3=Severe and 4 = incapacitating
Effectiveness of PUR0110 on inflammatory bowel disease questionnaire (IBDQ) score | At week 2
  Effectiveness of PUR0110 compared to placebo as per Change from baseline in inflammatory bowel disease questionnaire (IBDQ) score.
Effectiveness of PUR0110 on proportion of subjects with treatment failure defined as unchanged, worsened or missing modified Mayo score | At week 2
  Effectiveness of PUR0110 compared to placebo as per : Proportion of subjects with treatment failure;
Effect of PUR0110 on biomarkers of inflammation | At week 2
  Change from baseline in exploratory biomarkers - serum IL-2, IL-6, IL8, IFN-γ, TNF-α, TGF-β, IL-4, IL-10, IL-17, IL-23, hβD-2, MDA, LXA4, GSH and LTB4 levels in serum and biopsies; plasma and urinary isoprostane levels and serum lipoxin A4 levels..
Effect of PUR0110 on C-reactive Protein (CRP), high sensitivity CRP (hsCRP), erythrocyte sedimentation rate (ESR), Fecal Falprotectin (FCP) and Fecal Lactoferrin (FL) compared to placebo | At week 2
  Change from baseline in CRP, hs-CRP, ESR, FCP and FL .
Effect of PUR0110 on M30 apoptosome in serum and biopsies | At week 2
  Effect of PUR0110 on M30 apoptosome in serum and biopsies compared to placebo
Effect of PUR0110 on M65 apoptosome in serum and biopsies | At week 2
  Effect of PUR0110 on M65 apoptosome in serum and biopsies compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Theophilus J Gana, MD, PhD, Study Director — Devonian Health Group Inc.; Michael Rünzi, Prof. Dr. med., Principal Investigator — Essen-Werden, Germany
Locations (6):
- Germany (6):
  - PurGenesis Investigational Site, Jena
  - PurGenesis Investigational Site, Köln-Merheim
  - PurGenesis Investigational Site, Ludwigshafen
  - PurGenesis Investigational Site, Minden
  - PurGenesis Investigational Site, Oelde
  - PurGenesis Investigational Site, Werden